CLINICAL TRIAL: NCT03067883
Title: Evaluation of Efficacy and Safety of Ombitasvir, Paritaprevir, and Ritonavir Plus Ribavirin Based Therapy for Chronic Hepatitis C With or Without Compensated Cirrhosis in Haemodialysis Patients
Brief Title: Efficacy and Safety of Qurevo Plus Ribavirin Based Therapy for Hepatitis C With or Without Cirrhosis in Haemodialysis Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Mohamed Naguib Abdelmen'em Mohamed, Principle Investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Master (No 142)
Record Dates: First submitted 2017-01-23; First posted 2017-03-01 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ombitasvir; paritaprevir; Ritonavir

STUDY DESIGN:
Intervention Model Description: Prospective, cohort, open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (1):
- interventional Qurevo group (Experimental): A total of 40 HCV treatment naïve patients with or without compensated cirrhosis on regular hemodialysis will be enrolled in the study.
  * These patients will receive intervention of '25 mg ombitasvir, 150 mg paritaprevir, and 100 mg ritonavir' (2 capsules Qurevo®) plus ribavirin 200 mg daily for 12 weeks.
  * Qurevo will be given once daily (on the day of dialysis, it will be given after dialysis session).
  * Ribavirin will be given once daily (on the day of dialysis, it will be given 4 hrs before dialysis session ).
  Interventions: Drug: Ombitasvir, Paritaprevir and Ritonavir

INTERVENTIONS:
Drug: Ombitasvir, Paritaprevir and Ritonavir — A total of 40 HCV treatment naïve patients with or without compensated cirrhosis on regular hemodialysis will be enrolled in the study.
  * These patients will receive an intervention of '25 mg ombitasvir, 150 mg paritaprevir, and 100 mg ritonavir' (2 capsules Qurevo®) plus ribavirin 200 mg daily for 12 weeks.
  * Qurevo will be given once daily (on the day of dialysis, it will be given after dialysis session).
  * Ribavirin will be given once daily (on the day of dialysis, it will be given 4 hrs before dialysis session ).
  Other Names: qurevo

SUMMARY:
To evaluate efficacy and safety of Ombitasvir, paritaprevir, and ritonavir plus ribavirin based therapy for chronic hepatitis C with or without compensated cirrhosis in haemodialysis patients.

DETAILED DESCRIPTION:
The aim of this study is;

To evaluate the efficacy and safety of ombitasvir, paritaprevir, and ritonavir based therapy for chronic hepatitis C with or without compensated cirrhosis in HCV treatment naïve patients receiving long-term haemodialysis through assessment of:

1. The proportion of patients with a sustained virological response (HCV RNA <25 IU/mL) 12 weeks after the last dose of study drug (SVR12).
2. To determine withdrawal rate related to side effects and /or adverse effects for patients receiving at least 1 dose of the study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Under regular HD for at least 6 months
2. Clinically stable condition as outpatients.
3. Treatment naïve patients with serum positive for HCV GT4 with HCV RNA > 1000 IU/ml by PCR.
4. White blood cell count > 2500/mm^3.
5. Platelet count > 7500/mm^3.
6. Patients categorised as having compensated cirrhosis had a diagnosis of cirrhosis based on a previous screening liver FibroTest score of 0·72 or lower (eg, Metavir Fibrosis Score >3 [including 3/4 or 3-4] ).

Exclusion Criteria:

1. Confirmed pregnancy.
2. HCV-HIV co infection.
3. HBV-HCV co infection.
4. Uncontrolled hyper or hypothyroidism.
5. For patients without cirrhosis, Patients will be excluded if alanine or aspartate aminotransferase more than five times the upper limit of normal, for patients with cirrhosis they will be excluded if alanine or aspartate aminotransferase are higher than seven times the upper limit of normal
6. Patients on peritoneal dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11-09 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response | After 12 weeks after the last dose
  The proportion of patients with a sustained virological response (HCV RNA <25 IU/mL) 12 weeks after the last dose of study drug (SVR12).

SECONDARY OUTCOMES:
Treatment related withdrawal rate | during treatment period, average duration 3 months
  To determine withdrawal rate related to side effects and /or adverse effects for patients receiving at least 1 dose of the study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Mai Mohamed Naguib Abd Elmen'em, B.pharm, Principal Investigator — Ain Shams University
Locations (1):
- Maadi armed forces hospital, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided